CLINICAL TRIAL: NCT04174092
Title: Catastrophism in Chronic Inflammatory Rheumatism
Acronym: CRIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL 2019/CGV/01; 2019.A01715-52 (Other: ANSM)
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Chronic Inflammatory Rheumatism
Keywords: Catastrophism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rheumatoid arthritis (Experimental): Filling in several self-questionnaires: on function (HAQ), pain EVA, quality of life (SF12, EQ5D), anxiety score (GAD-7), insomnia score (ISI), catastrophic score (PCS), coping score (coping ability, CSQ), compliance scores (CQR, Health Insurance Compliance Assessment Questionnaire) and fibromyalgia diagnostic score (FiRST), activity of rheumatic disease (RAID, RAPID-3) Patients will be seen at 3, 6 and 12 months
  Interventions: Other: completing self-questionnaires
- spondyloarthritis (Experimental): Filling in several self-questionnaires: on function (HAQ), pain EVA, quality of life (SF12, EQ5D), anxiety score (GAD-7), insomnia score (ISI), catastrophic score (PCS), coping score (coping ability, CSQ), compliance scores (CQR, Health Insurance Compliance Assessment Questionnaire) and fibromyalgia diagnostic score (FiRST), activity of rheumatic disease (BASDAI, BASFI).
  Patients will be seen at 3, 6 and 12 months
  Interventions: Other: completing self-questionnaires
- Psoriatic arthritis (Experimental): Filling in several self-questionnaires: on function (HAQ), pain EVA, quality of life (SF12, EQ5D), anxiety score (GAD-7), insomnia score (ISI), catastrophic score (PCS), coping score (coping ability, CSQ), compliance scores (CQR, Health Insurance Compliance Assessment Questionnaire) and fibromyalgia diagnostic score (FiRST), activity of rheumatic disease (BASDAI, BASFI).
  Patients will be seen at 3, 6 and 12 months
  Interventions: Other: completing self-questionnaires

INTERVENTIONS:
Other: completing self-questionnaires — completing self-questionnaires on quality of life, anxiety, insomnia, activity of rheumatic disease and catastrophism

SUMMARY:
Catastrophic is defined as a negative cognitive and emotional response based on inadequate pain expression. It has three components: rumination, amplification and vulnerability. The assessment of catastrophism is carried out using a validated questionnaire called the "Pain Catatrophizing Scale" (PCS).

Recent studies highlight the significant impact of catastrophism in neuromuscular and mechanical rheumatic diseases such as gonarthrosis gonalgia and low back pain. In these diseases, it has been shown that catastrophism has a negative impact both on the experience of pain and on the response to different types of treatments (medical and surgical). Several studies have implemented multidisciplinary management and in particular cognitive-behavioural therapy with an improvement in the pain experience in patients who are catastrophic.

In chronic inflammatory rheumatic diseases such as rheumatoid arthritis, spondyloarthritis and psoriatic arthritis, the prevalence and impact of catastrophism is still poorly understood.

ELIGIBILITY:
Inclusion Criteria:

* Major patients, hospital follow-up, with RA according to ACR 2010 criteria, or spondyloarthritis according to ASAS 2009 criteria or according to AMOR or psoriatic arthritis according to Caspar 2006 criteria.
* Patient who has given free and informed consent.
* Patient who has signed the consent form.
* Patient affiliated or benefiting from a health insurance plan.
* Adult patient (≥18 years old).

Exclusion Criteria:

* Patient under the protection of justice, under guardianship or curatorship.
* Patient unable to express consent.
* Patient for whom it is impossible to provide informed information.
* Poor command and understanding of the French language making it impossible to complete self-questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2022-12-17 (Actual)

PRIMARY OUTCOMES:
catastrophic assessment | Day 0
  Pain Catastrophism Scale (0= no catastrophism, 52 = maximum catastrophism)
catastrophic assessment | at 3 months
  Pain Catastrophism Scale (0= no catastrophism, 52 = maximum catastrophism)
catastrophic assessment | at 6 months
  Pain Catastrophism Scale (0= no catastrophism, 52 = maximum catastrophism)
catastrophic assessment | at 12 months
  Pain Catastrophism Scale (0= no catastrophism, 52 = maximum catastrophism)

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (2):
- France (2):
  - CHU de Montpellier, Montpellier
  - CHU de Nîmes, Nîmes